CLINICAL TRIAL: NCT00877383
Title: A Randomized, Double-blind, Controlled, Parallel-group, 12-week Study to Compare the Efficacy and Safety of the Combination of Indacaterol 150 µg Once Daily With Open Label Tiotropium 18 µg Once Daily Versus Open Label Tiotropium 18 µg Once Daily in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Indacaterol Plus Tiotropium Versus Tiotropium Alone in Patients With Chronic Obstructive Pulmonary Disease
Acronym: INTRUST2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2351
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; COPD; indacaterol; tiotropium; bronchodilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol 150 μg and tiotropium 18 μg (Experimental): Patients inhaled indacaterol 150 μg and tiotropium 18 μg once daily in the morning between 8:00 AM and 11:00 AM for 12 weeks. Indacaterol was delivered blinded via a single-dose dry-powder inhaler (SDDPI). Tiotropium was delivered open-label via the manufacturer's proprietary inhalation device (HandiHaler®). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Tiotropium 18 μg
- Tiotropium 18 μg (Active Comparator): Patients inhaled placebo to indacaterol 150 μg and tiotropium 18 μg once daily in the morning between 8:00 AM and 11:00 AM for 12 weeks. Placebo to indacaterol was delivered blinded via a single-dose dry-powder inhaler (SDDPI). Tiotropium was delivered open-label via the manufacturer's proprietary inhalation device (HandiHaler®). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Tiotropium 18 μg; Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Indacaterol 150 μg and tiotropium 18 μg
Drug: Tiotropium 18 μg — Tiotropium was supplied in powder filled capsules together with the manufacturer's proprietary inhalation device (HandiHaler®).
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Tiotropium 18 μg

SUMMARY:
This study assessed the efficacy and safety of indacaterol (150 µg once daily [od]) when combined with tiotropium (18 µg od) versus tiotropium (18 µg od) treatment alone in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2007) and:

  * Smoking history of at least 10 pack-years
  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) ≤ 65% and ≥ 30% of the predicted normal value
  * Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria:

* Patients who have received systemic corticosteroids and/or antibiotics and/or was hospitalized for a COPD exacerbation in the 6 weeks prior to screening or during the run-in period
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1142 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceticals, Study Director — Novartis Pharmaceuticals
Locations (166):
- United States (106):
  - Novartis Investigator Site, Anniston, Alabama
  - Novartis Investigator Site, Birmingham, Alabama
  - Novartis Investigator Site, Jasper, Alabama
  - Novartis Investigator Site, Mobile, Alabama
  - Novartis Investigator Site, Glendale, Arizona
  - Novartis Investigator Site, Phoenix, Arizona
  - Novartis Investigator Site, Scottsdale, Arizona
  - Novartis Investigator Site, Little Rock, Arkansas
  - Novartis Investigator Site, Buena Park, California
  - Novartis Investigator Site, Fullerton, California
  - Novartis Investigator Site, Mission Viejo, California
  - Novartis Investigator Site, San Ramon, California
  - Novartis Investigator Site, Santa Barbara, California
  - Novartis Investigator Site, Sepulveda, California
  - Novartis Investigator Site, Spring Valley, California
  - Novartis Investigator Site, Torrance, California
  - Novartis Investigator Site, Vista, California
  - Novartis Investigator Site, Boulder, Colorado
  - Novartis Investigator Site, Centennial, Colorado
  - Novartis Investigator Site, Colorado Springs, Colorado
  - Novartis Investigator Site, Denver, Colorado
  - Novartis Investigative Site, Glastonbury, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigator Site, Clearwater, Florida
  - Novartis Investigator Site, Destin, Florida
  - Novartis Investigator Site, Maitland, Florida
  - Novartis Investigator Site, Miami, Florida
  - Novartis Investigator Site, Miami Beach, Florida
  - Novartis Investigator Site, Ocala, Florida
  - Novartis Investigator Site, Pensacola, Florida
  - Novartis Investigator Site, Port Orange, Florida
  - Novartis Investigator Site, South Miami, Florida
  - Novartis Investigator Site, Tamarac, Florida
  - Novartis Investigator Site, Tampa, Florida
  - Novartis Investigator Site, Couer D'Alene, Idaho
  - Novartis Investigator Site, Downers Grove, Illinois
  - Novartis Investigator Site, Elk Grove Village, Illinois
  - Novartis Investigator Site, River Forest, Illinois
  - Novartis Investigator Site, Springfield, Illinois
  - Novartis Investigator Site, Shawnee, Kansas
  - Novartis Investigator Site, Crescent Springs, Kentucky
  - Novartis Investigator Site, Lexington, Kentucky
  - Novartis Investigator Site, Louisville, Kentucky
  - Novartis Investigator Site, Shreveport, Louisiana
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigator Site, Troy, Michigan
  - Novartis Investigator Site, Chaska, Minnesota
  - Novartis Investigator Site, Edina, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Rochester, Minnesota
  - Novartis Investigator Site, Saint Paul, Minnesota
  - Novartis Investigator Site, Columbia, Missouri
  - Novartis Investigator Site, Kansas City, Missouri
  - Novartis Investigator Site, Ozark, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Billings, Montana
  - Novartis Investigator Site, Kalispell, Montana
  - Novartis Investigator Site, Bellevue, Nebraska
  - Novartis Investigator Site, Lincoln, Nebraska
  - Novartis Investigator Site, Papillion, Nebraska
  - Novartis Investigator Site, Henderson, Nevada
  - Novartis Investigative Site, Brick, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Ocean City, New Jersey
  - Novartis Investigative Site, Bayside, New York
  - Novartis Investigative Site, Great Neck, New York
  - Novartis Investigative site, Larchmont, New York
  - Novartis Investigative Site, Burlington, North Carolina
  - Novartis Investigator Site, Charlotte, North Carolina
  - Novartis Investigative Center, Raleigh, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigator Site, Statesville, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigator Site, Fargo, North Dakota
  - Novartis Investigator Site, Grand Forks, North Dakota
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigator Site, Cincinnati, Ohio
  - Novartis Investigator Site, Cleveland, Ohio
  - Novartis Investigator Site, Toledo, Ohio
  - Novartis Investigator Site, Oklahoma City, Oklahoma
  - Novartis Investigator Site, Eugene, Oregon
  - Novartis Investigative Site, Allentown, Pennsylvania
  - Novartis Investigative Site, Beaver, Pennsylvania
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Phoenixville, Pennsylvania
  - Novartis Investigative Site, Pawtucket, Rhode Island
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigator Site, Charleston, South Carolina
  - Novartis Investigator Site, Easley, South Carolina
  - Novartis Investigator Site, Greenville, South Carolina
  - Novartis Investigator Site, North Charleston, South Carolina
  - Novartis Investigator Site, Spartanburg, South Carolina
  - Novartis Investigator Site, Union, South Carolina
  - Novartis Investigator Site, Dallas, Texas
  - Novartis Investigator Site, Fort Worth, Texas
  - Novartis Investigator Site, Houston, Texas
  - Novartis Investigator Site, Tyler, Texas
  - Novartis Investigator Site, Salt Lake City, Utah
  - Novartis Investigative Site, Abingdon, Virginia
  - Novartis Investigative Site, Fredericks, Virginia
  - Novartis Investigator Site, Renton, Washington
  - Novartis Investigator Site, Spokane, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
- Canada (12):
  - Novartis Investigator Site, Gatineau
  - Novartis Investigator Site, Joliette
  - Novartis Investigator Site, Mirabel
  - Novartis Investigator Site, Mississauga
  - Novartis Investigator Site, Montreal
  - Novartis Investigative Site, Québec
  - Novartis Investigator Site, Saint-Jérôme
  - Novartis Investigator Site, Sainte-Foy
  - Novartis Investigator Site, Sherbrooke
  - Novartis Investigator Site, Toronto
  - Novartis Investigator Site, Trois-Rivières
  - Novartis Investigator Site, Windsor
- Colombia (4):
  - Novartis Investigative Site, Armenia
  - Novartis Investigator Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigator Site, Cali
- Czechia (7):
  - Novartis Investigative Site, Karlovy Vary
  - Novartis Investigative Site, Kladno
  - Novartis Investigative Site, Kroměříž
  - Novartis Investigative SIte, Liberec
  - Novartis Investigative Site, Rokycany
  - Novartis Investigative Site, Strakonice
  - Novartis Investigative Site, Třebíč
- Hungary (4):
  - Novartis Investigative Site, Érd
  - Novartis Investigative Site, Füzesabony
  - Novartis Investigator Site, Győr
  - Novartis Investgative Site, Százhalombatta
- India (9):
  - Novartis Investigator Site, Ahmedabad
  - Novartis Investigator Site, Bangalore
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Indore
  - Novartis Investigative Site, Jaipur
  - Novartis Investigator Site, Ludhiana
  - Novartis Investigative Site, Panjim
  - Novartis Investigator Site, Trivandrum
- Netherlands (6):
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Helmond
  - Novartis Investigative Site, Veldhoven
  - Novartis Investigative Site, Zutphen
- Slovakia (8):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigator Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Štúrovo
- Spain (10):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Almería
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigator Site, Madrid
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigator Site, Pozuelo de Alarcón
  - Novartis Investigator Site, Riudecols
  - Novartis Investigative Site, San Boi de Llobregat
  - Novartis Investigator Site, Seville
  - Novartis Investigative Site, Vilassar de Mar

REFERENCES:
- [Derived] Mahler DA, D'Urzo A, Bateman ED, Ozkan SA, White T, Peckitt C, Lassen C, Kramer B; INTRUST-1 and INTRUST-2 study investigators. Concurrent use of indacaterol plus tiotropium in patients with COPD provides superior bronchodilation compared with tiotropium alone: a randomised, double-blind comparison. Thorax. 2012 Sep;67(9):781-8. doi: 10.1136/thoraxjnl-2011-201140. Epub 2012 Apr 27. PMID 22544891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Started | 572 | 570
Completed | 543 | 533
Not Completed | 29 | 37
Not completed — Adverse Event | 13 | 14
Not completed — Lost to Follow-up | 5 | 3
Not completed — Subject withdrew consent | 3 | 12
Not completed — Subject no longer requires study drug | 2 | 0
Not completed — Administrative problems | 2 | 0
Not completed — Protocol deviation | 2 | 6
Not completed — Unsatisfactory therapeutic effect | 1 | 0
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg | Total
Number analyzed (Participants) | 572 | 570 | 1142
Age Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.83) | 62.8 (8.98) | 62.9 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 183 | 395
  Male | 360 | 387 | 747

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 8 Hours Post-dose at the End of the Study (Week 12, Day 84)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, 4, 6, and 8 hours post-dose at the end of the study (Week 12, Day 84). The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 8 hours post-dose at the end of the study (Week 12, Day 84)
Population: Full analysis set (FAS): All randomized patients who received at least 1 dose of study drug, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 530 | 504
Liters | 1.46 (0.011) | 1.34 (0.011)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of the Study (Week 12 + 1 Day, Day 85)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of the study. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: End of the study (Week 12 + 1 day, Day 85)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 565 | 564
Liters | 1.34 (0.010) | 1.27 (0.010)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 8 Hours Post-dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, 4, 6, and 8 hours post-dose on Day 1. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 8 hours post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 551 | 540
Liters | 1.40 (0.007) | 1.33 (0.007)

4. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose on Day 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose on Day 2. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose on Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 563 | 558
Liters | 1.34 (0.008) | 1.26 (0.008)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, and 4 hours post-dose on Day 1. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 4 hours post-dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 556 | 550
Liters | 1.38 (0.007) | 1.32 (0.007)

6. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose at the End of the Study (Week 12, Day 84)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5 and 30 minutes; and 1, 2, 3, and 4 hours post-dose at the end of the study (Week 12, Day 84). The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: From 5 minutes to 4 hours post-dose at the end of the study (Week 12, Day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Number analyzed (Participants) | 532 | 511
Liters | 1.48 (0.011) | 1.34 (0.011)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Week 12)
Description: Safety population: All patients who received at least 1 dose of study drug.
Arm/Group | Indacaterol 150 μg and Tiotropium 18 μg | Tiotropium 18 μg
Serious Adverse Events (participants affected / at risk) | 19/572 | 18/570
Other Adverse Events (participants affected / at risk) | 83/572 | 70/570
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg and Tiotropium 18 μg (N=572) | Tiotropium 18 μg (N=570)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg and Tiotropium 18 μg (N=572) | Tiotropium 18 μg (N=570)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 38 | 52
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.